CLINICAL TRIAL: NCT02797457
Title: Medical Economic Evaluation of Bilateral Allograft of Hands and Forearms
Acronym: ARMEDIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL15_0084
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Bilateral Traumatic Amputation of Upper Limbs
Keywords: Bilateral amputation of the forearms; Bilateral allograft; Prosthetic forehands; Medical economic evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft (Other): Bilateral allograft of the hands and forearms.
  Interventions: Procedure: Bilateral allograft of the hands and forearms.
- Prostheses (Other): Prosthetic forehands
  Interventions: Procedure: Prosthetic forehands

INTERVENTIONS:
Procedure: Bilateral allograft of the hands and forearms. — Bilateral allograft of the hands and forearms.
  Arms: Allograft
Procedure: Prosthetic forehands — Prosthetic forehands
  Arms: Prostheses

SUMMARY:
The double amputation of the forearms is a rare handicap that seriously impacts the autonomy and the quality of life of patients, social and familial exclusion, and dependence on third parties for everyday activities.

The management of these patients is nearly exclusively through the use of prostheses. Certain patients refuse this solution, or remain penalized by the absence of sensitivity , the lack of precision in movements, and body image issues related to the amputation; the double graft of hands and forearms may, in this circumstance, be the only solution.

Since January 2000, date of the first double hand graft, six bilateral grafts of hands have been performed at the Hospices Civils de Lyon. This first study reported the feasibility of the graft. The functional results obtained after the double transplant have allowed patients to recover complete autonomy for everyday activities, at the price of an immunosuppressive treatment. We have found that these very good functional results are maintained over time and, for a certain number of patients, to return to work which is a factor of social integration.

The rate of medical complications (metabolic, infectious, oncological), essentially related to the immunosuppressive treatment, is not greater to that found for other types of graft, but are considered as a limiting factor for the development of this strategy. These results are confirmed by international experience that is of the same order. Only a few rare cases of re-amputation have been reported in patients for whom the immunosuppressive treatment was discontinued or following vascular thrombosis.

A new study is required to continue this evaluation and to compare double graft to prostheses in terms costs, quality of life, usefulness, satisfaction, autonomy, and social integration. The results of this study will allow the placement of these strategies in the management of patients with double amputation of the hands and forearms.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria common to the 2 groups of patients (allograft group and protheses group):

* Adult aged 18 to 60 years
* Double amputated of both forearms

Transplant eligibility criteria (for allograft group)

* Minimum interval between amputation and graft of three months (no maximal delay)
* Absence of previous psychiatric history contraindicating the graft and psychological maturity, according to two psychiatrists who have evaluated the patient
* No previous history of malignant tumor in remission for less than 5 years
* American Society of Anesthesiology (ASA) score ≤ 2
* New York Heart Association (NYHA) grade ≥ 1
* Creatinine clearance ≥ 60 ml/min/1.73m²
* Absence of badly controlled sever hypertension

Exclusion Criteria:

* Mono amputated patients
* Malignant tumor or previous history of malignant tumor for which the risk of recurrence at 5 years is greater than 5%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2031-10-16 (Estimated); Study Completion 2031-10-16 (Estimated)

PRIMARY OUTCOMES:
Treatment cost | 36 months
  Treatment cost of double amputated patients by bilateral allograft of the hands and forearms or by prostheses

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Serice de Rééducation et Réadaptation fonctionnelles - Centre Jacques Calvé - Fondation Hopale, Berck
  - Service de Médecine Physique et Réadapatation fonctionnelle - Centre de Médecine Physique et de Réadaptation La Tour de Gassies, Bruges
  - Serice de Médecine Physique et Réadaptation - Hôpital d'Instruction des Armées Percy, Clamart
  - Serice de Rééducation et Réadaptation fonctionnelles - Centre l'Espoir, Lille
  - Serice de Médecine Physique et Réadaptation des patients amputés - Centre Médico-Chirugical et de Réadaptation des Massues, Lyon
  - Service de Chirurgie de la Transplantation - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - Serice de Rééducation et Réadaptation fonctionnelles - Centre Médical de Rééducation Romans Ferrari, Miribel
  - Service de Médecine Physique et Réadaptation - Institut Régional de Médecine Physique et de Réadaptation, Nancy
  - Serice de Rééducation fonctionnelle - Centre Mutualiste de Rééducation et Réadaptation fonctionnelles de Kerpape, Ploemeur
  - Serice de Rééducation et Réadaptation fonctionnelles - Hôpital Henry-Gabrielle - Hospices Civils de Lyon, Saint-Genis-Laval
  - Service de Rééducation et appareillage - Institut Robert Merle d'Aubigné, Valenton